CLINICAL TRIAL: NCT05347836
Title: Monocyte Soluble Activation Markers sCD14 and sCD163 in Children With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Maher Mokhtar Ahmed, Doctor, Assiut University
Other Study IDs: Monocyte activation markers
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children diagnosed to have T1DM with a minimum duration of five years
  Interventions: Diagnostic Test: ELISA
- Healthy children
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Determination of serum levels of sCD14 and sCD163 using ELISA

SUMMARY:
The study aims to compare serum levels of sCD14 and sCD163 in children with type 1 Diabetes Mellitus with healthy controls, study the distribution of monocyte subsets in children with T1DM , correlate monocyte subsets and their soluble activation markers sCD14 and sCD163 with parameters reflecting islet β-cell insufficiency in children with T1DM.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is T-cell mediated autoimmune disease in which the function of insulin-secreting pancreatic β-cells is impaired due to autoreactive immune cell-mediated destruction (insulitis). Although adaptive immunity has always been the focus for scientists in studying the pathogenesis of T1DM, yet, innate immunity also plays a critical role. Alterations in innate immune responses drive autoimmune pathogenesis, with involvement in the initial break in tolerance and the later failure of regulation. Several studies suggest that the development of T1DM is strongly associated with different immune cells, including monocytes. Specifically, an increase in the monocyte population has been shown to trigger β-cell destruction during insulitis. Intermediate monocytes may serve as M2 macrophage precursors with high anti-inflammatory properties, producing IL-10. However, other studies reported them to have an antigen-presenting function with a dendritic cell-like feature. Upon antigen stimulation, they became the main producers of inflammatory factors, like TNF-α which has been shown to correlate with the severity of T1DM. Activation of circulating monocytes to a pro-inflammatory state induces the shedding of membrane bound CD14 (mCD14) to soluble CD14. Compared to other acute phase proteins, sCD14 was found to be the most sensitive in T1DM. Soluble CD163 is present in blood serum as a result of shedding the CD163 membrane form of activated monocyte-macrophage-lineage cells in the course of inflammation. Plasma sCD163 is widely used as an immunomodulator with anti-inflammatory properties. It was found to be increased in T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Children of any age and sex diagnosed with T1DM (according to WHO criteria) with a minimum duration of five years will be included.

Exclusion Criteria:

* Children with other with coexisting autoimmune, chronic, and acute inflammatory diseases.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with type 1 Diabetes Mellitus Pediatric Endocrinology Unit in Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
To compare the levels of monocyte soluble activation markers among children with T1DM and healthy controls | Baseline
  To compare the levels of sCD14 and sCD163 among children with T1DM and healthy controls using ELISA

REFERENCES:
- [Background] Ismail NA, Abd El Baky AN, Ragab S, Hamed M, Hashish MA, Shehata A. Monocyte chemoattractant protein 1 and macrophage migration inhibitory factor in children with type 1 diabetes. J Pediatr Endocrinol Metab. 2016 Jun 1;29(6):641-5. doi: 10.1515/jpem-2015-0340. PMID 27054595
- [Background] Morgan NG, Leete P, Foulis AK, Richardson SJ. Islet inflammation in human type 1 diabetes mellitus. IUBMB Life. 2014 Nov;66(11):723-34. doi: 10.1002/iub.1330. Epub 2014 Dec 11. PMID 25504835
- [Background] Kim TK, Lee MS. Innate immune receptors in type 1 diabetes: the relationship to cell death-associated inflammation. Biochem Soc Trans. 2020 Jun 30;48(3):1213-1225. doi: 10.1042/BST20200131. PMID 32510139
- [Background] Marshak-Rothstein A. Autoimmunity--promoting and stabilizing innate immunity 'UNWUCHT'. Immunol Rev. 2016 Jan;269(1):7-10. doi: 10.1111/imr.12387. No abstract available. PMID 26683141
- [Background] Mysliwska J, Smardzewski M, Marek-Trzonkowska N, Mysliwiec M, Raczynska K. Expansion of CD14+CD16+ monocytes producing TNF-alpha in complication-free diabetes type 1 juvenile onset patients. Cytokine. 2012 Oct;60(1):309-17. doi: 10.1016/j.cyto.2012.03.010. Epub 2012 Apr 7. PMID 22484242
- [Background] Ancuta P, Weiss L, Haeffner-Cavaillon N. CD14+CD16++ cells derived in vitro from peripheral blood monocytes exhibit phenotypic and functional dendritic cell-like characteristics. Eur J Immunol. 2000 Jul;30(7):1872-83. doi: 10.1002/1521-4141(200007)30:73.0.CO;2-2. PMID 10940876
- [Background] Wong KL, Tai JJ, Wong WC, Han H, Sem X, Yeap WH, Kourilsky P, Wong SC. Gene expression profiling reveals the defining features of the classical, intermediate, and nonclassical human monocyte subsets. Blood. 2011 Aug 4;118(5):e16-31. doi: 10.1182/blood-2010-12-326355. Epub 2011 Jun 7. PMID 21653326
- [Background] Harms RZ, Ostlund KR, Cabrera MS, Edwards E, Fisher M, Sarvetnick N. Confirmation and Identification of Biomarkers Implicating Environmental Triggers in the Pathogenesis of Type 1 Diabetes. Front Immunol. 2020 Sep 15;11:1922. doi: 10.3389/fimmu.2020.01922. eCollection 2020. PMID 33042112
- [Background] Laursen TL, Wong GL, Kazankov K, Sandahl T, Moller HJ, Hamilton-Dutoit S, George J, Chan HL, Gronbaek H. Soluble CD163 and mannose receptor associate with chronic hepatitis B activity and fibrosis and decline with treatment. J Gastroenterol Hepatol. 2018 Feb;33(2):484-491. doi: 10.1111/jgh.13849. PMID 28618015
- [Background] Llaurado G, Gonzalez-Clemente JM, Maymo-Masip E, Subias D, Vendrell J, Chacon MR. Serum levels of TWEAK and scavenger receptor CD163 in type 1 diabetes mellitus: relationship with cardiovascular risk factors. a case-control study. PLoS One. 2012;7(8):e43919. doi: 10.1371/journal.pone.0043919. Epub 2012 Aug 24. PMID 22937125
- [Background] Ratajczak W, Atkinson SD, Kelly C. The TWEAK/Fn14/CD163 axis-implications for metabolic disease. Rev Endocr Metab Disord. 2022 Jun;23(3):449-462. doi: 10.1007/s11154-021-09688-4. Epub 2021 Sep 20. PMID 34542797
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34542797/
- Available data/document: Study Protocol — https://www.degruyter.com/document/doi/10.1515/jpem-2015-0340/html